CLINICAL TRIAL: NCT06779370
Title: Evaluation of the Effect of Calcium Silicate-Based Root Canal Medicament on Antifungal-Antibacterial Activity and Post-Operative Pain After Retreatment
Brief Title: Effect of Calcium Silicate-Based Root Canal Medicament After Retreatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Meltem Sümbüllü, Assistant Professor Dr. Meltem Sümbüllü, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14244
Record Dates: First submitted 2025-01-12; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Antibacterial Agents; Postoperative Dental Pain; Antifungal Agents
Keywords: calcium silicate based root canal medicament; calcium hydroxide based root canal medicament; bacterial load; antibacterial effect; antifungal effect; postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — calcium silicate; Calcium Hydroxide

STUDY DESIGN:
Intervention Model Description: two groups: group 1 calcium hydroxide based medicament (control group) group 2: calcium silicate based medicament
Who Masked: Outcomes Assessor
Masking Description: outcome assessments have performed by a investigator who was blinded to groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- calcium silicate based medicament (Experimental): Root canal lengths were determined using an electronic apex locator and a 15-K file. R25 Reciproc files were used at working lengths to remove the root canal filling. During instrumentation, the root canals were irrigated with saline solution. To obtain the first samples, three sterile paper points were placed at working length and the samples were transferred to an Eppendorf tube containing distilled water.
  Subsequently, the root canals were chemomechanically prepared, final irrigation activation was performed, and the second samples were collected in the same manner. The calcium silicate-based root canal medicament was placed in the canals, and the teeth were sealed with temporary fillings. A form was provided to assess the patients' postoperative pain levels over one week.
  At the second appointment, the medicament was removed, and third samples were collected using paper points with the same technique to evaluate antibacterial and antifungal effects. The root canal treatments of
  Interventions: Drug: Calcium Silicate
- calcium hydroxide based medicament (Active Comparator): Root canal lengths were determined using an electronic apex locator and a 15-K file. R25 Reciproc files were used at working lengths to remove the root canal filling. During instrumentation, the root canals were irrigated with saline solution. To obtain the first samples, three sterile paper points were placed at working length and the samples were transferred to an Eppendorf tube containing distilled water.
  Subsequently, the root canals were chemomechanically prepared, final irrigation activation was performed, and the second samples were collected in the same manner. The calcium hydroxide based root canal medicament was placed in the canals, and the teeth were sealed with temporary fillings. A form was provided to assess the patients' postoperative pain levels over one week.
  At the second appointment, the medicament was removed, and third samples were collected using paper points with the same technique to evaluate antibacterial and antifungal effects. The root canal treatments of
  Interventions: Drug: Calcium hydroxide

INTERVENTIONS:
Drug: Calcium Silicate — Root canal filling was removed with endodontic file. Sterile paper points were placed at working length to assess antibacterial and antifungal effects before the medicament was placed. Subsequently, the root canals were chemomechanically prepared, final irrigation activation was performed, and second samples were collected in the same manner. The calcium silicate-based root canal medicament was placed in the canals, and the teeth were sealed with temporary fillings. A form was provided to evaluate the patients' postoperative pain levels over one week. At the second appointment, the medicament was removed, and third samples were collected to assess antibacterial effects. The root canal treatments of the patients were completed. The antibacterial and antifungal effects of the medicaments were evaluated using PCR, and the patients' postoperative pain levels were recorded using follow-up forms.
  Other Names: calcium silicate based medicament group
  Arms: calcium silicate based medicament
Drug: Calcium hydroxide — Root canal filling was removed with endodontic file. Sterile paper points were placed at working length to assess antibacterial and antifungal effects before the medicament was placed. Subsequently, the root canals were chemomechanically prepared, final irrigation activation was performed, and second samples were collected in the same manner. The calcium hydroxide-based root canal medicament was placed in the canals, and the teeth were sealed with temporary fillings. A form was provided to evaluate the patients' postoperative pain levels over one week. At the second appointment, the medicament was removed, and third samples were collected to assess antibacterial effects. The root canal treatments of the patients were completed. The antibacterial and antifungal effects of the medicaments were evaluated using PCR, and the patients' postoperative pain levels were recorded using follow-up forms.
  Arms: calcium hydroxide based medicament

SUMMARY:
Calcium hydroxide is generally preferred in endodontics as an intracanal medicament due to its antimicrobial and biological effects. However, the antimicrobial effect of calcium hydroxide is limited. A new calcium silicate-based root canal medicament has been developed as an alternative to calcium hydroxide-based medicaments.

The aim of this study was to investigate the effects of calcium silicate-based root canal medicament on antibacterial, antifungal activity, and postoperative pain in root canal-treated teeth with periapical lesions.

DETAILED DESCRIPTION:
Sixty patients were randomly divided into two groups using a web-based program according to the selected medicament (calcium silicate-based root canal medicament or calcium hydroxide-based root canal medicament).

After the removal of gutta-percha from the root canals, the first samples were collected using paper points to evaluate antibacterial and antifungal effects. The root canals were then chemomechanically prepared, followed by final irrigation activation, and the second samples were collected. The selected root canal medicament was placed in the canals, and the patients were given a form to record their postoperative pain levels over one week.

At the second appointment, the medicaments were removed, and third samples were collected using paper points to assess antibacterial and antifungal effects. The root canal treatments of the patients were then completed. The antibacterial and antifungal effects of the medicaments were evaluated using PCR, and the patients' postoperative pain levels were recorded using follow-up forms.

ELIGIBILITY:
Inclusion Criteria:

* healthy patients with aged between 18-60.
* Incisor, canine, and premolar teeth that had previously undergone root canal treatment
* Incisor, canine, and premolar teeth with a diagnosis of chronic apical abscess or asymptomatic apical periodontitis
* teeth with only 1 root canal
* the patients had not used any antibiotics for 3 months before treatment

Exclusion Criteria:

* the presence of a root fracture
* teeth with any swelling
* ankyloses,
* periodontal pockets deeper than 4 mm.
* teeth which a rubber dam could not be performed
* patients with allergy to ibuprofen or ciprofloxacin were also excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-12 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
preoperative and postoperative levels of bacterial loud | one week
  The amounts of antibacterial loud was measured using a PCR kit.
preoperative and postoperative levels of antifungal loud | one week
  The amounts of antifungal loud was measured using a PCR kit.
postoperative pain levels | one week
  postoperative pain levels will be describe using the visual analog scale (VAS). The VAS was classified using the following scale [15]: no pain (0); mild pain (1-3); moderate pain (4-6), and severe pain (7-10).

CONTACTS AND LOCATIONS:
Overall Officials: meltem SÜMBÜLLÜ, DDS, Principal Investigator — Ataturk University
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mentes I, Sumbullu M. Effect of tricalcium silicate-based intracanal dressing on antibacterial-antifungal activity and postoperative pain intensity after non-surgical endodontic retreatment: randomized controlled clinical trial. Head Face Med. 2025 Nov 21;21(1):78. doi: 10.1186/s13005-025-00559-w. PMID 41272686